CLINICAL TRIAL: NCT06532019
Title: Randomized Multicenter Clinical Trial in Heart Failure Patients With Preserved Ejection Fraction (HFpEF) at Intermediate and High Risk of All-cause Death
Brief Title: Clinical Study of Active Intervention in High-risk HFpEF Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangtan Central Hospital (Other)
Collaborators: The First People's Hospital of Xiangtan City (Unknown); The Xiangtan People's Hospital (Unknown); The Xiangxiang People's Hospital (Unknown)
Responsible Party: Principal Investigator, Jianping Zeng, Dean, Xiangtan Central Hospital ,Director of cardiovascular clinic, Clinical Professor, Xiangtan Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HFpEF intervention trial
Record Dates: First submitted 2024-07-27; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: all-cause mortality

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care group (No Intervention): Patients in this group will receive usual medical care for heart failure.
- targeted intervention group (Experimental): Patients in this group, besides usal medical care for heart failure, will receive targeted therapy: correct hypoalbuminemia, anemia or hyponatremia, and try to enhance medication to lower NT-proBNP, CRP, NYHA Classification, to add diuretics for patients with higher RADs, multidiscipline intervention for patients complicating COPD, and actively reperfusion for ischemic HFpEF patients.
  Interventions: Other: Targeted intervention based on risk factors

INTERVENTIONS:
Other: Targeted intervention based on risk factors — Correct hypoalbuminemia, anemia or hyponatremia, and try to enhance medication to lower NT-proBNP, CRP, NYHA Classification, to add diuretics for patients with higher RADs, multidiscipline intervention for patients complicating COPD, and actively reperfusion for ischemic HFpEF patients.
  Arms: targeted intervention group

SUMMARY:
Based on inclusion and exclusion criteria, this experiment plans to include 924 Heart Failure with Preserved Ejection Fraction(HFpEF) patients with increased risk of all-cause death. The enrolled patients will divided into usual care group (n=462) and targeted intervention group (n=462) in a 1:1 ratio. The usual care patients will receive routine heart failure treatment. Patients in targeted intervention group, on top of routine therapy for heart failure, will receive further therapy targeting therapy to correct hypoalbuminemia, anemia or hyponatremia, and try to enhance medication to lower N-terminal pro brain natriuretic peptide (NT-proBNP), C-reactive protein(CRP), New York Heart Association(NYHA )Classification, to add diuretics for patients with higher right ventricular diameters(RADs),multidiscipline intervention for patients complicating chronic obstructive pulmonary disease(COPD), and actively reperfusion for ischemic HFpEF patients. The incidence of all-cause death will be compared after 3 years follow-up.The primary endpoint is the occurrence of all-cause mortality events during the follow-up period.

DETAILED DESCRIPTION:
Our newly finished study developed and validated a risk prediction model for all-cause mortality in patients with HFpEF based on real-world data. The nomogram prediction model included factors such as NT-proBNP, albumin, age, NYHA class III-IV, CRP, RADs, hemoglobin, COPD, hyponatremia, and Percutaneous Coronary Intervention(PCI). Discharged HFpEF patients with scores ≥200.37 were found to be associated with increased risk of all-cause death up to 3 years. In this trial, we sought to evaluate the impact of targeted risk factors intervention post-discharge in patients with with scores ≥200.37 on all-cause death up to 3 years.

Based on inclusion and exclusion criteria,We will enroll 924 patients with HFpEF and scores ≥200.37. The enrolled patients will divided into a usual care group (n=462) and targeted intervention group (n=462) in a 1:1 ratio. The usual care group patients will receive routine heart failure treatment, Patients in targeted intervention group, on top of routine therapy for heart failure, will receive further therapy targeting therapy to correct hypoalbuminemia, anemia or hyponatremia, and try to enhance medication to lower NT-proBNP, CRP, NYHA Classification, to add diuretics for patients with higher RADs, multidiscipline intervention for patients complicating COPD, and actively reperfusion for ischemic HFpEF patients. The primary endpoint is the occurrence of all-cause mortality events during the 3 years follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Discharged HFpEF patients with risk score > or equal 200.37.

Exclusion Criteria:

* Patients with a life expectancy of less than 1-year due to malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | The patients will be followed up for 3 years after they were enrolled.
  follow-up by clinical visit, telephone call or community visit

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xia, PH.D, Study Chair — Xiangtan Central Hospital

IPD SHARING:
Plan to Share IPD: No